CLINICAL TRIAL: NCT06979050
Title: Evaluation of the Ronnie Gardiner Method in Individuals With Stroke in Late Phase of Recovery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Karlstad University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-01269-01
Record Dates: First submitted 2025-05-06; First posted 2025-05-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Music-based intervention; Stroke rehabilitation; Ronnie Gardiner Method
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation. Neither participants nor intervention providers will be masked due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music-based intervention (Experimental): Participants randomized to the intervention group will receive the Ronnie Gardiner Method (RGM), a rhythm- and music-based training program, in group sessions led by a certified instructor. The intervention consists of 60-minute sessions, twice per week, for 12 consecutive weeks. The training incorporates coordinated movements, speech, and rhythm using visual symbols representing limbs and directions, performed to music with varying tempo and complexity. Exercises are designed to improve motor function, balance, coordination, and cognitive engagement. Sessions are conducted primarily in standing to optimize balance effects.
  Interventions: Behavioral: The Ronnie Gardiner Method
- Waiting-list (No Intervention): Waiting list, receiving the same intervention after the final follow-up assessment three months post-intervention.

INTERVENTIONS:
Behavioral: The Ronnie Gardiner Method — The intervention involves participants performing coordinated movements while saying specific cue words, synchronized to rhythmic music. The exercises are guided by a visual notation system consisting of 19 colored symbols that represent different body parts and movements. Red symbols indicate movements on the left side of the body, while blue symbols represent the right side. Each symbol corresponds to a specific movement and verbal cue. Exercises are typically performed standing to maximize balance effects and are accompanied by rhythmic, often popular, music to enhance engagement and motivation. Complexity can be increased by adjusting the tempo of the music or combining multiple symbols. Training sessions are conducted in groups, led by certified instructors, twice per week for 12 weeks (60 minutes per session), with an additional home-based practice session each week.
  Other Names: RGM
  Arms: Music-based intervention

SUMMARY:
Stroke is a common condition that often leads to long-term disabilities, significantly affecting individuals' quality of life and imposing substantial societal costs. There is growing evidence that physical rehabilitation can improve motor function, well-being, and quality of life even in the chronic phase after stroke. In recent years, rhythm- and music-based interventions have gained increasing attention as promising tools in neurorehabilitation. The Ronnie Gardiner Method (RGM) is a structured, music-based training method that engages motor, sensory, cognitive, and emotional functions simultaneously. While preliminary studies have shown positive effects of RGM in individuals with Parkinson's disease, there is limited research on its impact in stroke rehabilitation, particularly in the chronic phase.

This randomized controlled multicenter study aims to evaluate the effects of RGM training in individuals aged 18 and older who are more than six months post-stroke. Participants will be randomly assigned to either an intervention group receiving RGM training twice per week for 12 weeks, or to a passive control group. The primary outcome is balance, assessed by the Mini-BESTest. Secondary outcomes include gait, upper limb function, cognitive abilities such as working memory and divided attention, and health-related quality of life. Additionally, qualitative data will be collected to explore participants' and trainers' experiences regarding motivation, engagement, and perceived impact on daily participation. The study is expected to provide valuable evidence on the clinical usefulness of RGM in chronic stroke rehabilitation and its potential to be implemented as part of community-based, cost-effective rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling individuals with stroke that occurred > 6 months ago
* Cognitive ability corresponding to at least 25 out of 30 points on the Montreal Cognitive Assessment (MoCA)
* Functional disability corresponding to a Modified Rankin Scale (mRS) score of 2-3
* No assistance required for daily activities during participation (e.g., can independently travel to measurement/training sites and use the restroom)
* Ability to stand for 2 minutes without support and walk 10 meters with or without assistive devices, but without supervision

Exclusion Criteria:

* Severe visual and/or hearing impairments that would interfere with study participation
* Participation in regular sessions with RGM after August 2024
* Previous experience playing a musical instrument (defined as practicing >1 hour/week in the past 10 years)
* A score of less than 25 on the Montreal Cognitive Assessment (MoCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Balance performance measured by the Mini Balance Evaluation Systems Test (Mini-BESTest) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The mini-BESTest (Mini Balance Evaluation Systems Test) is a shortened version of the BESTest, designed to assess balance and functional mobility, especially in individuals with neurological or musculoskeletal conditions. It focuses on balance deficits across domains like postural control, gait, stability, and anticipatory responses. With 14 items compared to the original 36, the mini-BESTest is quicker to administer, making it more practical for clinical use. It evaluates four main balance systems:
  * Anticipatory Postural Adjustments: Preparing and adjusting posture for movements.
  * Reactive Postural Control: Responding to unexpected balance challenges.
  * Sensory Orientation: Using sensory input (like vision and proprioception) for balance.
  * Dynamic Gait: Stability and efficiency while walking, including maintaining balance during movement.
  Minimum score is 0 points, maximum score is 28 points. Higher scores indicate better balance control.

SECONDARY OUTCOMES:
Concern about falling measured by the Falls Efficacy Scale-International (FES-I) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  FES-I is a tool used to assess a person's confidence in performing daily activities without falling. It consists of 16 questions that cover a range of activities, from walking and bathing to social interactions. The scale helps identify individuals who may have a fear of falling, which can impact their participation in everyday life.
  Minimum score is 16 points, maximum score is 64 points. A higher score indicates greater concern about falling, and it's commonly used in older adults or individuals at risk of falls to guide interventions aimed at improving balance and reducing fall risk.
Working memory measured by the Memory Test (Immediate and Delayed Recall) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The test assesses the ability to recall a read text immediately after it is read aloud and after a few minutes, when another test is conducted (delayed recall).
Cognitive flexibility and inhibitory control measured by the Victoria Stroop Test | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  Measures cognitive flexibility, attention, and response inhibition. It involves naming the color of printed words that may or may not match the color they describe, requiring the individual to suppress automatic reading responses. The test is commonly used to assess executive function, particularly in individuals with neurological conditions. It includes three conditions, and outcomes include reaction time and number of errors. Higher interference scores indicate poorer inhibitory control.
Visuospatial memory and organization measured by the Rey-Osterrieth Complex Figure Test | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The Rey-Osterrieth Complex Figure Test is a neuropsychological assessment used to evaluate visuospatial abilities, memory, attention, and executive function. Individuals are asked to copy a complex geometric figure and later reproduce it from memory after a delay. It is commonly used to assess cognitive impairments in various neurological conditions. Scoring is based on accuracy and placement of figure components. Higher scores indicate better visuospatial memory and organizational performance.
Physical performance measured by the Short Physical Performance Battery (SPPB) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  A clinical tool used to assess lower extremity function and mobility in older adults. It includes tests of balance, gait speed, and chair stands to evaluate physical performance. The SPPB is commonly used to predict disability, falls, and overall functional decline.
  Minimal score is 0 points, maximum score is 12 points. Higher score indicates better physical function.
Functional mobility and gait performance measured by the 10-Meter Walk Test (10MWT) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The 10-Meter Walk Test (10MWT) is a quick assessment used to measure walking speed over 10 meters at the individual's self-selected pace. It evaluates functional mobility, gait efficiency, and balance. The test is commonly used to monitor progress and predict functional outcomes in people with neurological or musculoskeletal conditions.
Physical capacity including aerobic capacity and endurance measured by the 6-Minute Walk Test (6MWT) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The 6-Minute Walk Test (6MWT) measures the distance an individual can walk at a self-paced speed over six minutes. It assesses aerobic capacity, endurance, and functional mobility. The test is widely used to evaluate cardiovascular and pulmonary function in clinical and rehabilitation settings. The test measures the distance a person can walk in six minutes on a flat, hard surface, typically a 30-meter course.
Upper extremity function measured by The Observational Drinking Task Assessment | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The Observational Drinking Task Assessment is used to evaluate upper limb function, motor control, and coordination during a simulated drinking task. The individual is observed while reaching for, grasping, and bringing a cup to the mouth. It is often used in neurological rehabilitation to assess functional use of the affected arm.
  Minimal score is 0 points, maximal score is 15 points. Higher scores indicate worse outcome, i.e., more impairments in the upper extremity.
Finger dexterity and fine motor skills measures by the 9-Hole Peg Test (9HPT) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The 9-Hole Peg Test is a standard assessment used to measure finger dexterity and fine motor skills. The individual is required to place and remove pegs from a pegboard as quickly as possible. It is commonly used to assess hand function in individuals with neurological conditions, such as multiple sclerosis or stroke.
Health-related quality of life and functional recovery after a stroke measured by the Stroke Impact Scale 16 (SIS-16) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The Stroke Impact Scale 16 (SIS-16) is a self-reported questionnaire used to assess the health-related quality of life and functional recovery after a stroke. It consists of 16 items that measure various aspects of physical, emotional, and social functioning. The scale helps track recovery progress and guide rehabilitation in stroke survivors.
  Minimal score is 16 points, and maximum is 80. Higher score indicates a better function and lower impact on everyday life.
Severity of depressive symptoms measured by the Montgomery-Åsberg Depression Rating Scale (MADRS) | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-administered assessment used to evaluate the severity of depressive symptoms. It consists of 10 items that assess mood, sleep, appetite, and other emotional and physical symptoms associated with depression. The MADRS is commonly used in clinical settings to monitor treatment progress and assess depression severity.
  Minumum score is 0 points, and maximum score is 60. Higher scores indicate more severe symptoms of depression.
General health-realted quality of life measured by the Research and development (RAND) 36-item health survey | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The RAND-36 is a health survey used to assess an individual's overall health-related quality of life. It consists of 36 items that measure eight domains, including physical functioning, emotional well-being, social functioning, and general health perceptions. The RAND-36 is widely used in both clinical and research settings to evaluate health outcomes across various conditions.
  Minimal score is 0 points, maximal score is 100 points. Higher values indicate better self-reported health-related quality of life.
Cost-effectiveness evaluated with the standardized European Quality of Life (EuroQol) questionnaire with 5 dimensions | At baseline, at 12 weeks (end of intervention), and at 24 weeks (3-month follow-up)
  The EuroQol 5D 5L (EQ-5D-5L) is a standardized instrument used to assess health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated on five levels of severity. The EQ-5D-5L is commonly used in clinical trials, healthcare evaluations, and to measure the impact of treatments on patients' well-being.
  Minimal score is 0 on a visual analogue scale, and 100 is maximum. A higher score indicates better health in general. Scores is used to evaluate an interventions cost-effectiveness.

OTHER OUTCOMES:
Various cognitive domains measured by the Montreal Cognitive Assessment (MoCA) | Only at baseline
  The Montreal Cognitive Assessment (MoCA) is a screening tool used to assess cognitive function and detect mild cognitive impairment. It evaluates various cognitive domains, including memory, attention, language, visuospatial skills, and executive function. The MoCA is commonly used in clinical settings to identify early signs of cognitive decline, such as in Alzheimer's disease or other neurodegenerative conditions. In our study, it will be used as an inclusion criterion.
  Minimal score is 0 points, maximum score is 30 points. In our study, a score of 25 is required to be included in the study. The MoCA is only used as a screening tool at baseline.
Participants' enjoyment of the interventions measured by the Physical Activity Enjoyment Scale (PACES) | After 12 weeks of treatment
  The Physical Activity Enjoyment Scale (PACES) is a tool used to assess an individual's enjoyment of physical activity. It consists of several18 items that measure positive and negative feelings associated with engaging in physical exercise. PACES is commonly used in research and clinical settings to understand motivation and promote long-term adherence to physical activity.
  Minimal score is 18 points, and maximum score is 126 points. Higher score indicates higher enjoyment of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Pohl, PhD, Principal Investigator — Göteborg University
Locations (3):
- Sweden (3):
  - Folkuniversitetet, Gothenburg
  - Resurscentrum, Karlstad
  - Neurologiska rehabiliteringskliniken, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, data will be prepared and made available in accordance with Swedish data protection reulations and the University of Gothenburg's Rules for Research Data Management. In line with these regulations, data containing personal information will be deposited in the Swedish National Data Service repository under a "restricted access" model.
  Under this model, a description of the data (metadata) together with relevant documentation files will be openly published, while the actual data files will not be directly accessible. Researchers wishing to access the data must submit a request through the repository, and each request will be reviewed before access is granted.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Ghai S, Pohl P. Evaluation of the Ronnie Gardiner Method in individuals with stroke in the late phase of recovery: a protocol for a single-blind multicentre randomised controlled trial. BMJ Open. 2026 Feb 4;16(2):e107178. doi: 10.1136/bmjopen-2025-107178. PMID 41638729
- See also: Related Info — https://www.gu.se/forskning/rehabilitering-med-rytm-och-musik-en-studie-av-ronnie-gardiner-method-vid-stroke